CLINICAL TRIAL: NCT05291351
Title: Comparison of the Impacts of Pea, Lentil, and Oat Flour Particle Size on Postprandial Glycemic Response and Appetite in Healthy Adults
Brief Title: Impact of Pea, Lentil and Oat Flour Particle Size on Glycemic Response in Healthy Adults
Acronym: PLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University of Saskatchewan (Other); Saskatchewan Food Industry Development Center (Unknown)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 20180182
Record Dates: First submitted 2022-02-28; First posted 2022-03-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition; Diabetes; Malnutrition; Protein; Obesity
Keywords: Nutrition; Glycemic response; Protein quality; Food processing
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus; Kwashiorkor; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, crossover acute trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pea (Experimental): Treatment 1: crackers made with 25% whole pea flour + 75% all-purpose wheat flour; Treatment 2: crackers made with 25% coarse pea flour + 75% all-purpose wheat flour; Treatment 3: crackers made with 25% fine pea flour + 75% all-purpose wheat flour; Treatment 4: crackers made with 100% all-purpose wheat flour (control)
  Interventions: Other: Crackers made with whole, coarse, or fine pea and/or wheat flour
- Lentil (Experimental): Treatment 1: crackers made with 25% whole lentil flour + 75% all-purpose wheat flour; Treatment 2: crackers made with 25% coarse lentil flour + 75% all-purpose wheat flour; Treatment 3: crackers made with 25% fine lentil flour + 75% all-purpose wheat flour; Treatment 4: crackers made with 100% all-purpose wheat flour (control)
  Interventions: Other: Crackers made with whole, coarse, or fine lentil and/or wheat flour
- Oats (Experimental): Treatment 1: porridge made with whole oat flour; Treatment 2: porridge made with coarse oat flour; Treatment 3: porridge made with fine oat flour; Treatment 4: porridge made with commercial oat flour (control)
  Interventions: Other: Porridge made with oat flour

INTERVENTIONS:
Other: Crackers made with whole, coarse, or fine pea and/or wheat flour — Participants will consume 1 of the 4 treatments at each of 4 study sessions in random orders such that by the end of the study, they will have consumed all 4 treatments. They will be given 10 minutes to consume the entire treatment with a glass of water.
  Arms: Pea
Other: Crackers made with whole, coarse, or fine lentil and/or wheat flour — Participants will consume 1 of the 4 treatments at each of 4 study sessions in random orders such that by the end of the study, they will have consumed all 4 treatments. They will be given 10 minutes to consume the entire treatment with a glass of water.
  Arms: Lentil
Other: Porridge made with oat flour — Participants will consume 1 of the 4 treatments at each of 4 study sessions in random orders such that by the end of the study, they will have consumed all 4 treatments. They will be given 10 minutes to consume the entire treatment with a glass of water.
  Arms: Oats

SUMMARY:
The study looks at the comparative effects of food products made with pea, lentil, and oat flour of various particle sizes on postprandial glycemic response, appetite and food intake, and amino acid release in healthy adults.

DETAILED DESCRIPTION:
A total of 60 participants (30 males, 30 females) will take part in this study at the University of Toronto. Twenty participants will be recruited to each one of three trials (pea, lentil or oat) and will attend 4 study sessions where they will consume crackers/porridge made with pea, lentil, oat, or wheat flours of different particle sizes. Questionnaires will be filled out to assess their recent food intake, physical activity, sleep quality, stress level, appetite, physical comfort, and energy/fatigue level, as well as tastefulness of the food. Blood samples will be collected at fasting and at various time points over a 2 hour period after eating to measure blood glucose, insulin, and amino acid concentrations. Before leaving, participants will receive an all-you-can-eat pizza meal to assess their food intake.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* BMI 18.5-29.9 kg/m2
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to maintain current dietary supplement use throughout the trial.
* Willing to abstain from alcohol consumption for 24h prior to all test visits.
* Willing to avoid vigorous physical activity for 24h prior to all test visits.
* Understanding the study procedure and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Smoking
* Thyroid problems
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, a malabsorptive syndrome, pancreatitis, gallbladder or biliary disease.
* Presence of a gastrointestinal disorder or surgeries within the past year.
* Known to be pregnant or lactating.
* Unwillingness or inability to comply with the experimental procedures and to follow our safety guidelines.
* Allergies to peanuts and nuts.
* Known intolerances, sensitivity or allergy to any ingredients in the study products: pea flour, lentil flour, oat flour and whole wheat flour.
* Regular breakfast skipping (consumes breakfast less than 5 days a week)
* Extreme dietary habits (i.e Atkins diet, very high protein diets, etc.) or restrained eaters, identified by a score of ≥ 11 on the Eating Habits Questionnaire
* Uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg) as defined by the average blood pressure measured at screening.
* Weight gain or loss of at least 10lbs in previous three months.
* Excessive alcohol intake (more than 2 drinks per day or more than 9 drinks per week).
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose or that could affect the outcome of the study as per investigator's judgment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in postprandial glycemic response | Blood glucose will be measured at baseline and at 15, 30, 45, 60, 90, 120, and 140 minutes after treatment consumption. Insulin will be measured at baseline and every half an hour after treatment consumption over 2 hours.
  Blood collection via finger prick to analyze blood glucose (glucometer reading) and serum insulin concentration (μIU/mL).

SECONDARY OUTCOMES:
Subjective appetite | At baseline and at 15, 30, 45, 60, 90, 120, and 140 minutes after treatment consumption.
  Motivation to Eat Adaptive Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Food intake | 2 hours after treatment consumption.
  Measured via amount of pizza (g) consumed at an ad libitum pizza meal.
Protein quality | At baseline and every half hour after treatment consumption over a period of 2 hours, and after pizza meal.
  Intravenous blood collection to analyze amino acid concentrations (μmol/L) to determine amino acid release.
Physical comfort | At baseline and at 15, 30, 45, 60, 90, 120, and 140 minutes after treatment consumption.
  Physical Comfort Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Energy & fatigue | At baseline and at 15, 30, 45, 60, 90, 120, and 140 minutes after treatment consumption.
  Energy and Fatigue Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.
Treatment palatability | Immediately after treatment consumption.
  Treatment Palatability Visual Analogue Scales measured based on a score between 0 to 100. A higher score indicates higher outcome.

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou CZC, Anderson GH, Fan W, Vien S, Ai Y, Tulbek M, Fabek H. Increasing particle size of oat flours decreases postprandial glycemia and increases appetite in healthy adults. Nutr Res. 2024 Oct;130:81-94. doi: 10.1016/j.nutres.2024.07.006. Epub 2024 Jul 25. PMID 39366276